CLINICAL TRIAL: NCT06196814
Title: Efficay and Satety of PD-1/VEGR Bispecific Antibodies (AK112) Plus Platinum-based Chemotherapy for EGFR/ALK/ROS1 Positve NSCLC: A Multiple Centers, Multiple Cohorts, Dose Escalation Phase II Apple Study
Brief Title: AK112 Plus Platinum-based Chemotherapy for EGFR/ALK/ROS1 Positve NSCLC
Acronym: Apple
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Prof., Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCH20231225
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Efficacy

STUDY DESIGN:
Intervention Model Description: This study will be devided into three cohorts. Cohort A for EGFR mutation NSCLC, Patient with NGS idenfied EGFR sensitive mutation NSCLC who failed from first line Osimertinib will be included. The 3+3 stud will conducted for dose escalation for AK112 （from 20mg to 30mg), and than the fix dose will be set up for cohort A, B and C.
  Cohort B for ALK fusion NSCLC, Patient with NGS idenfied ALK fusion NSCLC who failed from first line Alectinib will be included. All the patients will be devided two group,3'ALK and 3'ALK with reteintion of 5'ALK. All the patients will be treated with PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy.
  Cohort C for ROS1 fusion NSCLC, Patient with NGS idenfied ROS1 fusion NSCLC who failed from first line crizotinib or Entrectinib will be included. All the patients will be treated with PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy.
  We will colect the satety and efficacy data for all the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort of EGFR Sensitve Mutant NSCLC (Experimental): Efficay, Satety and Dose Escalation of AK112 plus Platinum-based Chemotherapy for EGFR Sensitive mutant NSCLC who Failed from First-Line Osimertinib.
  Interventions: Drug: PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy
- Cohort of ALK Fusion NSCLC (Experimental): Efficay and Satety of PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy for ALK fusion NSCLC who Failed from First-Line Osimertinib.
  Interventions: Drug: PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy
- Cohort of ROS1 Fusion NSCLC (Experimental): Efficay and Satety of PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy for ROS1 fusion NSCLC who Failed from First-Line Crizotinib.
  Interventions: Drug: PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy

INTERVENTIONS:
Drug: PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy — PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy.

SUMMARY:
The investigators want to evaluated the Efficay and Satety of PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy for EGFR/ALK/ROS1 Positve NSCLC who Failed from First-Line Standard Treatment.

DETAILED DESCRIPTION:
The investigators want to evaluated the Efficay and Satety of PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy for EGFR/ALK/ROS1 Positve NSCLC who Failed from First-Line Standard Treatment.

This study will be devided into three cohorts. Cohort A for EGFR mutation NSCLC, Patient with NGS idenfied EGFR sensitive mutation NSCLC who failed from first line Osimertinib will be included. The 3+3 stud will conducted for dose escalation for AK112 （from 20mg to 30mg), and than the fix dose will be set up for cohort A, B and C.

Cohort B for ALK fusion NSCLC, Patient with NGS idenfied ALK fusion NSCLC who failed from first line Alectinib will be included. All the patients will be devided two group,3'ALK and 3'ALK with reteintion of 5'ALK. All the patients will be treated with PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy.

Cohort C for ROS1 fusion NSCLC, Patient with NGS idenfied ROS1 fusion NSCLC who failed from first line crizotinib or Entrectinib will be included. All the patients will be treated with PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy.

The investigators will collect the satety and efficacy data for all the patients.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects selected for this study must meet all of the following criteria:

  1. Sign written informed consent before implementing any trial-related procedures;
  2. Age ≥18 years old and ≤75 years old;
  3. No limit on the gender;
  4. The ECOG score is 0 or 1.
* The investigators want to evaluated the Efficay and Satety of PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy for EGFR/ALK/ROS1 Positve NSCLC who Failed from First-Line Standard Treatment.

This study will be devided into three cohorts.

* Cohort A for EGFR mutation NSCLC, Patient with NGS idenfied EGFR sensitive mutation NSCLC who failed from first line Osimertinib will be included. The 3+3 stud will conducted for dose escalation for AK112 （from 20mg to 30mg), and than the fix dose will be set up for cohort A, B and C.
* Cohort B for ALK fusion NSCLC, Patient with NGS idenfied ALK fusion NSCLC who failed from first line Alectinib will be included. All the patients will be devided two group,3'ALK and 3'ALK with reteintion of 5'ALK. All the patients will be treated with PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy.
* Cohort C for ROS1 fusion NSCLC, Patient with NGS idenfied ROS1 fusion NSCLC who failed from first line crizotinib or Entrectinib will be included. All the patients will be treated with PD-1/VEGR bispecific antibodies (AK112) plus Platinum-based Chemotherapy.

The investigators will collect the satety and efficacy data for all the patients.

Exclusion Criteria:

* Histological or cytological pathology confirmed the presence of a small cell carcinoma component, or a squamous cell carcinoma as a major component
* Patients who have received immunotherapy previously, including immune checkpoint inhibitors (such as anti-PD-1/L1, anti-CTLA-4 , anti-LAG-3, etc.), immune checkpoint activators (such as ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), immune cell therapy and any other treatment targeting the immunity mechanism.
* Previously received other anti-tumor therapy for advanced stages of NSCLC (stages IIIB to IV) (including cytotoxic chemotherapy used with radiotherapy, systemic chemotherapy, and anti-VEGFR therapy) .

Patients who have previously undergone adjuvant/neoadjuvant chemotherapy with the aim of curing non-metastatic diseases are eligible for inclusion in this study if disease progression occurs at least 6 months after the completion of the last chemotherapy cycle.

* Concurrent enrollment in another clinical trial is allowed, unless it involves a non-interventional clinical study or the follow-up period of an interventional study (defined as the time elapsed from the initiation of the first drug to at least 4 weeks after the last drug administration in the previous clinical study or beyond 5 half-lives of the investigational drug in that study, whichever is shorter).
* Received TKI treatment within the 2 weeks preceding the first dose; underwent palliative local therapy for non-target lesions within the 2 weeks preceding the first dose; received non-specific immunomodulatory therapy within the 2 weeks preceding the first dose, such as interleukins, interferons, thymosin alpha-1, tumor necrosis factor, etc. (excluding IL-11 used for treating thrombocytopenia); received herbal medicine or traditional Chinese medicine with anti-tumor indications within the 1 week preceding the first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
RP2D | 2 months
  We want to evaluate the best dose for treatment.
ORR | 12 months
  Overall response rate
PFS | 12 months
  Progression free survival time

IPD SHARING:
Plan to Share IPD: No